CLINICAL TRIAL: NCT04869332
Title: A Prospective Randomised Controlled Clinical Trial: Three Cancellous Screws Versus Four Cancellous Screws for Fixation of Femoral Neck Fractures
Brief Title: Three Cancellous Screws Versus Four Cancellous Screws for Femoral Neck Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUTH LY MCS
Record Dates: First submitted 2021-04-09; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Femoral Neck Fractures; Internal Fixation
Keywords: femoral neck fractures; multiple cancellous screws; RCT
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three-screw group (Active Comparator): three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck
  Interventions: Device: three cancellous screws
- four-screw group (Experimental): the fourth screw will be implanted in the horizontal direction of the femoral distance on the basis of the three screws.
  Interventions: Device: four cancellous screws

INTERVENTIONS:
Device: three cancellous screws — All patients with femoral neck fractures will be randomly divided into 2 groups at a ratio of 1:1. Three screws for internal fixation in the three-screw group, and three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck.
  Arms: three-screw group
Device: four cancellous screws — All patients with femoral neck fractures will be randomly divided into 2 groups at a ratio of 1:1. Four screws for internal fixation in the four-screw group, and the fourth screw will be implanted in the horizontal direction of the femoral distance on the basis of the three screws.
  Arms: four-screw group

SUMMARY:
This study is a prospective randomized controlled clinical study. Patients with femoral neck fracture (AO classification 31-B) will be randomly divided into three-screw fixation group and four-screw fixation group. The internal fixation failure rate (IFFR) and functional outcomes of the two groups will be compared and the patients will be followed up to 2 years after surgery.

DETAILED DESCRIPTION:
This is a prospective randomized controlled clinical trial. All patients will be randomly divided into 2 groups at a ratio of 1:1. The investigators will use three screws for internal fixation in the first group, and four screws for internal fixation in the second group. The relevant parameters of the sample calculation are α = 0.05 (one-sided) and β = 0.2. PASS 15 was used for calculation, and the final sample size was 290, 145 for each group. Subjects who meet all the inclusion conditions but do not meet any exclusion conditions and have signed the informed consent will be randomized, and each patient will be assigned a unique patient identification number, which will be used throughout the study. Using a computer random allocation system, eligible patients were randomly divided into the two groups at a ratio of 1:1. The investigators will perform preoperative preparations, intraoperative operations, and internal fixation in accordance with the instructions provided in the internal plant product packaging. The investigators only plan to include cases in which closed reduction can be successfully performed, so the investigators will exclude cases that require open reduction. For the three-screw group, three cancellous screws with an inverted triangle pattern are used to fix the fracture of femoral neck. For the four-screw group, the fourth screw will be implanted in the horizontal direction of the femoral distance on the basis of the three screws. After the operation, the subjects will be managed according to the standard nursing and rehabilitation procedures at the experimental site and the results of laboratory examinations will be recorded. Regular follow-up evaluations will be carried out after the operation until the end of the two-year follow-up or the end of the study. In this study, the internal fixation failure rate (IFFR) will be used as the main research endpoint, which is defined as the total incidence of cutouts, fractures. The results of the radiographic examination, the lateral X-ray film and computed tomography(CT), will be evaluated by an independent radiologist to determine whether there are cut-out or fracture of the internal plant. Secondary endpoints include: 1. Bone nonunion after 36 weeks: evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, it is defined as nonunion if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months. 2. Garden classification proportion, and Garden index for reduction assessment. 3. Clinical prognosis: o A 12-Item Short-Form Health Survey (SF-12) o Harris hip score. 4. Operation time, from the incision to internal fixation implanted. 5. The times of intraoperative fluoroscopy, average 25 milliseconds per X-ray shot, record the number of X-ray shot. 6. Postoperative adverse events within 2 years, including ipsilateral femoral head avascular necrosis, infection, wound hematoma, ipsilateral coxa vara, and ipsilateral limb shortening. In this study, it is difficult to blind anyone to randomization. However, considering that most of the patients may not have medical expertise, if the researchers do not inform them, the patients are the only people who may be blind. Investigators will try their best to reduce human-induced bias in experimental results. Investigators will use one-sided α = 0.05 for statistical tests and confidence interval calculations. P value <0.05 is considered statistically significant. SPSS (latest version: SPSS Inc., Chicago, IL, USA) will be used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with unilateral femoral neck fractures that will be treated with internal fixation
* According to AO fracture classification, subjects with the fracture type (31-B)
* Subjects (with the help of relatives) can understand the informed documents and patient questionnaires.
* Subjects (with the help of relatives) voluntarily provide written informed consent to participate in the clinical study and authorize the transfer of their information to the sponsor.
* The investigator believes that the subject can understand the clinical study, is willing and able to complete all research procedures and follow-up visits and can cooperate with the research procedures.
* In-label use of the MCS.

Exclusion Criteria:

* Subject does not provide voluntary consent to participate in the study.
* The researcher believes that the subjects have conditions that affect the participation and follow-up of this study. (for example, the patient lives in a remote area or has difficulty in going back to the hospital for follow-up or does not cooperate with the medical guidance and suggestions of the surgeon.)
* The subjects were pregnant or lactating women.
* The researchers believe that the subjects have psychological disorders, which may affect the treatment outcome.
* Garden classification III and IV of femoral neck fracture patients older than 65 years
* Concurrent hip osteoarthritis.
* Fractures where the operative treatment will occur more than three weeks after the primary injury
* Patients combined with femoral head fractures(31-C), femoral shaft fractures(32-A/B/C) or femoral trochanteric area fracture (31-A1/A2/A3).
* Pathological fracture (e.g., primary or metastatic tumor)
* Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined vascular injury, and combined osteofascial compartment syndrome
* Multiple systemic injuries judged by researchers not suitable for enrollment.
* Revision surgeries (for example, due to malunion, nonunion or infection)
* Concurrent medical conditions judged by researchers not suitable for enrollment, such as: metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc
* Patients with anaesthetic and surgical contraindications
* Patients known to be allergic to implant components
* Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
* Intemperance judged by researchers not suitable for enrollment (e.g., excessive daily drinking or smoking, drug abuse);
* Subjects participated in other clinical studies in the past 3 months, which may affect the outcome and follow-up according to the judgment of researchers.
* Subjects have significant neurological or musculoskeletal disorders or may have adverse effects on gait or weight-bearing (e.g., muscular dystrophy, multiple sclerosis, cerebral infarction, hemiplegia, Charcot arthropathy, avascular necrosis of the femoral head).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Internal fixation failure rate | from operation to 2-year follow-up after the surgery
  defined as the total incidence of internal plant cut-out and fracture

SECONDARY OUTCOMES:
Number of Participants with Bone nonunion | from operation to 9-month follow-up after the surgery
  evaluate bone healing according to the lateral X-ray examination. According to the regulations of Food and Drug Administration of the US, if there are no obvious signs of fracture healing 9 months after the fracture, or if there is no obvious difference in fracture space after three consecutive months, it is defined as nonunion.
Harris hip score | from operation to 2-year follow-up after the surgery
  the score value is from 0 to 100, and a higher score means a better outcome
operation time | intraoperative
  from the incision to internal fixation implanted.
The times of intraoperative fluoroscopy | intraoperative
  average 25 milliseconds per X-ray shot, record the number of X-ray shot
Garden index | from operation to 2-year follow-up after the surgery
  The fracture reduction will be considered unsatisfied if the index is less than 155 degrees or more than 180 degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Zhou, M.D., Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No